





## APPENDIX 6 - Consent form for semi-structured interviews

| raiticipant number | Particip | ant | number |
|--------------------|----------|-----|--------|
|--------------------|----------|-----|--------|

## **CONSENT FORM- Semi-Structured Patient and Professional Interviews (P-IGBC)**

**Title of project:** P-iGBC (Identification of **P**redictive factors of **I**ncidentally detected **G**all**B**ladder **C**ancer and prospective validation of a scoring system to allow selective histological analysis of the gallbladder)

Investigator(s): Mr. Somaiah Aroori, Mr Oliver Brown, Dr Lexy Sorrell, Prof. Jos Latour

| | If you agree please initial each statement as appropriate |
|---|---|
| 1. | I confirm that I have read the participant information sheet dated 06/09/2024 (version 2.1) for the interviews. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. |
| 3. | I understand that, to allow interviews to be arranged and for subsequent communication, personally identifiable information, including my name, email address, telephone number and/or home address will be shared with the research team and stored securely at University Hospitals Plymouth NHS Trust. |
| 4. | I understand that if I agree to participate in future research, the information collected about me in this study may be used to support other research in the future and may be shared anonymously with other researchers. |

IRAS number: 334671

FREIC 5550

Version 1.2 04 November 2024







| 5. | I understand that my data, in<br>during the interviews, may be<br>or dissertation), or published<br>would be anonymised, and i<br>(either directly or indirectly)<br>presentations or published s | pe used internally (for description of the control | or example, in a thesis<br>licly. However, my data<br>sible to identify me<br>nated reports, |
|---|---|---|---|
| 6. | 5. I understand that my de-identified data will be shared between University Hospitals Plymouth NHS Trust and the University of Plymouth for the purposes of analysis, and that it will contribute to a research degree being undertaken by one of the researchers. | | |
| 7. | 7. I understand that my privacy and confidentiality will be maintained at all stages of the study under the provisions of the Data Protection Act 2018. | | |
| 8. | . I understand that my interview will be audio and/or video recorded to gather all relevant information, and the recordings will be deleted immediately after transcription. | | |
| 9. | I agree to take part in the interviews. | | |
| 10. | 10. I would like to be sent a summary of the results of the research. I give permission for you to send this to me at my email address (optional, write email below): | | |
| Name | of Participant | Date | Signature |
| | of Person taking consent | Date | Signature |
| When | completed (Paper consent): copy for p | participant; original copy for | or researcher site file |

IRAS number: 334671

FREIC 5550

Version 1.2 04 November 2024

When completed (eConsent): emailed PDF copies for participant and for researcher site file